CLINICAL TRIAL: NCT06686108
Title: Safety and Efficacy Study of Demethylating Agents With Venetoclax in Preventing Recurrence of High-risk T-cell Lymphoblastic Lymphoma/Leukemia After Transplantation
Brief Title: Demethylating Agents Combined With Venetoclax for High-risk T-cell Lymphoblastic Lymphoma/Leukemia Post-Transplant Relapse Prevention
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHSYXY-T-LBL-AZA/VEN-Rel-2024
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-10

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION; Relapse
Keywords: T-cell lymphoblastic lymphoma/leukemia; relapse; allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Leukemia | interventions — Azacitidine; Decitabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- combination therapy (Experimental): There is only 1 arm. Combination therapy arm included venetoclax combined with hypomethylating agents such as azacitidine or decitabine. 1. venetoclax: 400mg/d, po, days 1-7 of each 28-day cycle. 2.For patients without TP53 mutation, azacitidine was administered: 32mg/m2/d, ih, days 1-5 of each 28-day cycle; for patients with TP53 mutation, decitabine was administered: 5mg/m2/d, iv, days 1-5 of each 28-day cycle.
  Interventions: Drug: Azacitidine (AZA) Days 1 - 5; Drug: Decitabine (DAC); Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine (AZA) Days 1 - 5 — Azacitidine, ih, 32mg/m2/d, days 1-5 of each 28-day cycle
Drug: Decitabine (DAC) — decitabine, 5mg/m2/d, days 1-5 of each 28-day cycle.
Drug: Venetoclax — venetoclax, 400mg/d, days 1-7 of each 28-day cycle

SUMMARY:
This study is a prospective, phase II clinical trial with the primary objective of assessing the effectiveness of demethylating agents combined with venetoclax in the prevention of recurrence after allogeneic hematopoietic stem cell transplantation (allo-HSCT) of high risk T-lymphoblastic lymphoma/leukemia (T-LBL/ALL) patients.

DETAILED DESCRIPTION:
The experimental group included high risk T-ALL/LBL patients after allo-HSCT, who received relapse prevention treatment with demethylating agents such as azacitidine or decitabine, combined with venetoclax.

The historical control consisted of high-risk T-ALL/LBL patients who received allo-HSCT but did not receive any prophylactic treatment from multiple centers, and their basic information, disease information, treatment details, and efficacy data were collected. Propensity score matching was conducted with historical data to compare the advantages and disadvantages of the experimental regimen with the control group.

The primary endpoint was the relapse-free survival(RFS) rate after prophylaxis, while secondary endpoints included cumulative incidence of relapse (CIR), overall survival (OS), and the GVHD-relapse-free survival (GRFS). This study aims to provide a effective and safer prophylaxis treatment for high-risk T-LBL/ALL patients after all-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* 1.14-55 years old, male,or female.
* 2.Patients with allo-HSCT due to T-LBL/ALL, the donor type is not limited.
* 3.ECOG score is 0-2 points.
* 4.Blood routine: ANC ≥ 1.0 × 109/L, PLT ≥ 50 × 109/L.
* 5.One of the following high-risk factors:
* a. Age of initial diagnosis ≥ 35 years old.
* b. Initial diagnosis of WBC ≥ 100 × 109/L.
* c. Initial diagnosis of LDH exceeding the upper limit of normal values.
* d. Initial diagnosis of bone marrow involvement (blast cells ≥ 5%).
* e. Initial diagnosis of a bulky in the mediastinum (longest diameter ≥ 10cm).
* f. ETP immunophenotype.
* g. During the induction chemotherapy process, 2 courses did not achieve partial remission and/or 4 courses did not achieve complete remission.
* h. Residual lesions before transplantation: Flow cytometry analysis showed that the proportion of abnormal lymphoid cells in the bone marrow was greater than 0.01%; Positive detection of minimal residual lesions in molecular biology; PET-CT scan shows that residual lesions are still active.
* i. Based on the ELN recommendation based on adult T-ALL: gene mutations involving myeloid related genes, RAS/PI3K/AKT, JAK/STAT signaling pathway, and epigenetics, such as FLT3, NRAS/KRAS, PTEN, IL7R, JAK1, JAK3, DNMT3A, IDH1, IDH2; TP53, BCL2 mutations; t (8; 14) (q24; q11)/MYC rearrangement; t (7; 19) (q34; p13)/TCR-LYL1，TCR-MEF2C; del(5q) (q14).
* j. High risk subgroups based on NGS definition: PI3K signaling pathway/NRAS, KRAS/TP53/IKZF1/DNTM3A/IDH1, IDH2 gene mutation with or without NOTCH1, FBXW7/PHF6/EP300 gene mutation.

Exclusion Criteria：

* 1.Central involvement during any course of the disease.
* 2.Patients who have not achieved complete remission before transplantation.
* 3.Identify those with available targeted drugs.
* 4.For those who are resistant to BCL-2 inhibitors before transplantation, if the disease progresses during the application process, or if 3-4 courses of induction therapy containing BCL2 inhibitors do not improve.
* 5.Individuals who are known to be allergic to demethylating drugs or venetoclax.
* 6.Individuals with grade 2 or more degrees of active acute GVHD.
* 7.Individuals with moderate to severe chronic GVHD.
* 8.T-LBL/ALL relapse (flow cytometry abnormal lymphocyte cell proportion>0.01%, WT1 positive, fusion gene positive, or extramedullary recurrence), or transplant rejection, bone marrow donor cell chimerism<95%.
* 9.Blood routine: ANC<1.0 × 109/L or PLT<50 × 109/L.
* 10.Combined with severe organ dysfunction; The ratio of aspartate aminotransferase (AST)/alanine aminotransferase (ALT) is more than 3 times the normal value or the normal value of direct bilirubin is more than 3 times; The endogenous creatinine clearance rate (Ccr) is less than 50mL/min or 1.5 times the normal value of blood creatinine, regardless of whether hemodialysis treatment is used.
* 11.Merge severe active infections.
* 12.Pregnant or lactating women.
* 13. Accepting other investigational drugs.
* 14.According to the researchers' assessment, the patient may have complications that could lead to other dangers.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
RFS | 1 year
  1-year relapse-free survival
RFS | 2 year
  2-year relapse-free survival

SECONDARY OUTCOMES:
CIR | 1 year
  1-year cumulative incidence of relapse
CIR | 2 year
  2-year cumulative incidence of relapse
OS | 1 year
  1-year overall survival
OS | 2 year
  2-year overall survival
GRFS | 1 year
  1-year graft-versus-host disease (GVHD)-free/relapse-free survival (GRFS) rates
GRFS | 2 year
  2-year graft-versus-host disease (GVHD)-free/relapse-free survival (GRFS) rates
cGVHD | 1 year
  1-year cumulative incidence of cGVHD
cGVHD | 2 year
  2-year cumulative incidence of cGVHD
adverse events | at the end of every cycle (each cycle is 28 days)
  adverse events during research

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided